CLINICAL TRIAL: NCT02301104
Title: A Phase 1, Open-label Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of TAS-102 in Patients With Advanced Solid Tumors and Varying Degrees of Hepatic Impairment.
Brief Title: A Phase I Study of TAS-102 in Patients With Advanced Solid Tumors With Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TO-TAS-102-106
Record Dates: First submitted 2014-11-13; First posted 2014-11-25 (Estimated); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Advanced Solid Tumors
Keywords: Liver Neoplasms; Hepatic; TAS-102; mCRC; Liver Impairment; Pharmacologic Actions; Liver Diseases; Liver; LFT; Advanced Solid Tumor; Pharmacokinetics
MeSH Terms: conditions — Liver Neoplasms; Liver Diseases | interventions — trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Mild Hepatic Impairment (Experimental): 35 mg/m2/dose of TAS-102 orally, twice daily on days 1-5 and days 8-12 of each 28-day cycle. Number of cycles: approximately 4 or until discontinuation criteria is met.
  Interventions: Drug: TAS-102
- Moderate Hepatic Impairment (Experimental): 35 mg/m2/dose of TAS-102 orally, twice daily on days 1-5 and days 8-12 of each 28-day cycle. Number of cycles: approximately 4 or until discontinuation criteria is met.
  Interventions: Drug: TAS-102
- Severe Hepatic Impairment (Experimental): 35 mg/m2/dose of TAS-102 orally, twice daily on days 1-5 and days 8-12 of each 28-day cycle. Number of cycles: approximately 4 or until discontinuation criteria is met.
  The dose level of severe cohort, if enrolled, will be determined based on the Interim Assessment of mild and moderate cohorts.
  Interventions: Drug: TAS-102
- Normal Hepatic Function (Experimental): 35 mg/m2/dose of TAS-102 orally, twice daily on days 1-5 and days 8-12 of each 28-day cycle. Number of cycles: approximately 4 or until discontinuation criteria is met.
  Interventions: Drug: TAS-102

INTERVENTIONS:
Drug: TAS-102

SUMMARY:
Study to evaluate the safety, tolerability, and pharmacokinetics of TAS-102 in patients with advanced solid tumors and varying degrees of hepatic impairment.

DETAILED DESCRIPTION:
This is a Phase 1, open-label study to evaluate the safety, tolerability, and pharmacokinetics of TAS-102 in patients with advanced solid tumors with varying degrees of hepatic impairment. The study is conducted in 2 parts: the Pharmacokinetic Part (Cycle 1) and the Extension Part (Cycles 2 and beyond). Patients may continue to receive treatment with TAS-102 during the study extension part only after completion of the Pharmacokinetic Part.

ELIGIBILITY:
Inclusion

1. Has provided written informed consent
2. Has advanced solid tumors (excluding breast cancer)
3. Has normal hepatic function, mild, moderate, or severe hepatic impairment
4. ECOG performance status of ≤2
5. Is able to take medications orally
6. Has adequate organ function
7. Women of childbearing potential must have a negative pregnancy test and must agree to adequate birth control if conception is possible. Males must agree to adequate birth control.

Exclusion

1. Certain serious illnesses or medical condition(s)
2. Has had certain other recent treatment e.g. major surgery, anticancer therapy, extended field radiation, received investigational agent, shunt in the liver within the specified time frames prior to study drug administration
3. Has received TAS-102
4. Has unresolved toxicity of greater than or equal to CTCAE Grade 2 attributed to any prior therapies
5. Is a pregnant or lactating female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
PK parameters of FTD, FTY, and TPI in plasma after a single dose of TAS-102 | Blood samples will be collected in Cycle 1 Day 1 and Day 12 at pre-dose, 0.5, 1, 2, 4, 6, 8, 10, and 12 hours post AM dose of TAS-102
  FTD, FTY and TPI: pharmacokinetic parameters Cmax, Tmax, AUC0-last, AUC0-inf, and T1/2. FTD and TPI: CL/F, Vd/F of TAS-102
Safety monitoring including adverse events, vital signs, and laboratory assessments | Through 30 days following last administration of study medication or until initiation of new anticancer treatment

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Mayo Clinic, Scottsdale, Arizona
  - Duarte Clinical Site, Duarte, California
  - Santa Monica Clinical Site, Santa Monica, California
  - Baltimore Clinical Site, Baltimore, Maryland
  - Boston Clinical Site, Boston, Massachusetts
  - Cleveland Clinical Site, Cleveland, Ohio
  - Pittsburgh Clinical Site, Pittsburgh, Pennsylvania
  - Dallas Clinical Site, Dallas, Texas